CLINICAL TRIAL: NCT00067587
Title: Prevalence of Morphologic and Metabolic Abnormalities in HIV Infected and Uninfected Young Women
Brief Title: Metabolic Abnormalities in HIV Infected and Uninfected Young Women
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 021
Record Dates: First submitted 2003-08-25; First posted 2003-08-26 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2016-02

CONDITIONS: HIV Infections; Hypercholesterolemia; Glucose Intolerance
Keywords: Treatment experienced; Treatment naive
MeSH Terms: conditions — HIV Infections; Hypercholesterolemia; Glucose Intolerance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- HIV Negative: HIV negative subjects
- HIV Positive - NEVER had ARV therapy.: HIV Positive - NEVER had ARV therapy.
- HIV positive, on a NNRTI, non-PI regimen: HIV positive, currently on a NNRTI, non-PI regimen for at least 3 months. Must NEVER have received a total of more than SIX months of PI-containing regimen and at least ONE year must have passed since receipt of last PI-containing regimen.
- HIV positive, on a PI, non-NNRTI regimen: HIV positive, currently on a PI, non-NNRTI regimen for at least 3 months. Must NEVER have received a total of more than SIX months of NNRTI-containing regimen and at least ONE year must have passed since receipt of last NNRTIcontaining regimen.
- HIV positive, on a non-PI, non-NNRTI: HIV positive, currently on a non-PI, non-NNRTI containing regimen for at least 3 months. Must NEVER have received a total of more than SIX months of PI- and/or NNRTI- containing regimen and at least ONE year must have passed since receipt of last PI- and/or NNRTI-containing regimen.

SUMMARY:
Though anti-HIV drugs can dramatically improve the health of people with HIV, some people taking these drugs develop serious long term effects in their metabolism. These effects include problems with bones, increased levels of blood sugar and lipids, and changes in body fat distribution. The purpose of this study is to see how many young women are experiencing these problems and how severe the problems are. This kind of study is the first step in determining how best to treat these problems.

DETAILED DESCRIPTION:
Patients on highly active antiretroviral therapy (HAART) regimens develop potentially deleterious metabolic effects, including insulin resistance, dyslipidemia, osteopenia and osteoporosis, and hyperlactatemia. Changes in body fat distribution and bone metabolism are also documented. There is considerable evidence that protease inhibitors (PI) can induce insulin resistance and increase triglyceride and cholesterol levels. It is now also clear that both metabolic changes and fat distribution abnormalities occur in PI-naive patients treated with nucleoside analogue reverse transcriptase inhibitors (NRTIs). In addition to class specific effects, there is emerging evidence that there are differences within each class of drug in the nature and magnitude of metabolic effects. This study will examine the metabolic effects of HAART in young women.

Adolescent women aged 12 through 24 years will be recruited into each of 5 treatment strata: Stratum 1 - HIV uninfected; Stratum 2 - HIV infected but never had HAART; Stratum 3 - HIV infected on NNRTI regimen for 3 or more months and less than 2 weeks of PI therapy; Stratum 4 - HIV infected on PI regimen for 3 or more months and less than 2 weeks of NNRTI therapy; and Stratum 5 - HIV infected on NRTI-only regimen for 3 or more months and less than 2 weeks of PI or NNRTI therapy. Participants in the study will have one study visit conducted over 1 or 2 days. The study visit will include survey questionnaires, DEXA scanning, anthropometric measurements, and blood tests examining lactate, glucose, and lipid metabolism.

ELIGIBILITY:
Inclusion criteria

* Negative serum or urine pregnancy test if not sterilized
* Tanner Stage 4 or 5
* Accessible medical and medication history
* Willing to fast and complete clinical and laboratory evaluations
* Willingness and ability to give consent or assent with parental permission

Exclusion criteria

* Refusal to fast for 8 hours prior to specimen collection
* Unable to obtain history
* Pregnancy in last 12 months or currently pregnant
* History of anorexia or bulimia
* Type I Diabetes mellitus
* Type II Diabetes mellitus and cannot omit medication for the 48 hour period prior to laboratory specimen collection

Ages: 12 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A total of up to 300 subjects may be enrolled in the study. The number of subjects in each study group will be as follow: 50 HIV negative subjects; 100 HIV positive subjects with no exposure to ART; and three groups of up to 50 HIV positive subjects each with different ART exposure histories.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2003-07; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Aldrovandi, MD, Study Chair — Children's Hospital Los Angeles
Locations (11):
- United States (11):
  - Children's Hopsital of Los Angeles, Los Angeles, California
  - University of California at San Diego, San Diego, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stoger Hospital of Cook County, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - Mt. Sinai Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- See also: Description of Adolescent Trials Network (ATN) and contact information — http://www.atnonline.org